CLINICAL TRIAL: NCT01009541
Title: An Open-Label, Multiple-Dose, Randomized, Crossover Study In Healthy Volunteers To Investigate The Pharmacokinetics Of Three Dose Strengths Of Pregabalin Controlled Release Formulations Administered Following An Evening Meal As Compared To The Immediate Release Formulation
Brief Title: An Investigation of the Absorption and Pharmacokinetics of Multiple Doses of Three Controlled Release Pregabalin Tablets as Compared to Multiple Doses of the Immediate Release Pregabalin Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081225
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2009-12

CONDITIONS: Healthy
Keywords: pregabalin pharmacokinetics bioavailability bioequivalence
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pregabalin controlled release, 82.5 mg (Experimental)
  Interventions: Drug: Pregabalin controlled release, 82.5 mg
- Pregabalin controlled release, 165 mg (Experimental)
  Interventions: Drug: Pregabalin controlled release, 165 mg
- Pregabalin controlled release, 330 mg (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg
- Pregabalin immediate release, 150 mg (Other): Reference Treatment
  Interventions: Drug: Pregabalin immediate release, 150 mg

INTERVENTIONS:
Drug: Pregabalin controlled release, 82.5 mg — 82.5 mg controlled release tablet administered once daily for three days.
  Arms: Pregabalin controlled release, 82.5 mg
Drug: Pregabalin controlled release, 165 mg — 165 mg controlled release tablet administered once daily for three days.
  Arms: Pregabalin controlled release, 165 mg
Drug: Pregabalin controlled release, 330 mg — 330 mg controlled release tablet administered once daily for three days.
  Arms: Pregabalin controlled release, 330 mg
Drug: Pregabalin immediate release, 150 mg — 150 mg immediate release capsules administered every 12 hours for three days
  Arms: Pregabalin immediate release, 150 mg

SUMMARY:
The purpose of this study is to 1) evaluate the extent of absorption of multiple doses of three pregabalin controlled release tablets as compared to multiple doses of the pregabalin immediate release capsule, 2) evaluate the pharmacokinetics of multiple doses of three pregabalin controlled release tablets as compared to multiple doses of pregabalin immediate release capsule and 3) evaluate the safety and tolerability of multiple doses of three pregabalin controlled release tablets as compared to multiple doses of the pregabalin immediate release capsule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve at steady-state for a dosing interval (AUCτ), Dose-adjusted AUCτ | 5 days
Minimum plasma concentration at steady-state within a dosing interval (Cmin) | 5 days
Maximum plasma concentration at steady-state (Cmax), time of Cmax at steady-state (tmax) | 5 days
The average plasma concentration at steady-state (Cav), half-life | 5 days
Peak:trough ratio at steady-state (PTR), peak to trough fluctuation at steady-state (PTF), and peak:trough swing at steady-state (PTS) | 5 days

SECONDARY OUTCOMES:
Safety endpoints include evaluation of adverse events. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081225&StudyName=An%20investigation%20of%20the%20absorption%20and%20pharmacokinetics%20of%20multiple%20doses%20of%20three%20controlled%20release%20pregabalin%20tablets%20as%20compared%20to%20